CLINICAL TRIAL: NCT01739101
Title: The Reproductive Life Plan in Midwifery Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Jenny Stern, RN, PhD-student, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UU-RLP-RCT-2012
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Delayed Childbearing; Pregnancy; Health Behavior; Lifestyle
MeSH Terms: conditions — Reproductive Behavior; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention group (Experimental): The intervention group answered a baseline questionnaire in the waiting room and received the intervention (Reproductive Life Plan) in addition to standard care.
  Interventions: Behavioral: Reproductive Life Plan
- Control group 1 (No Intervention): The control group 1 answered a baseline questionnaire in the waiting room and received standard care.
- Control group 2 (No Intervention): The control group 2 received standard care.

INTERVENTIONS:
Behavioral: Reproductive Life Plan — A structured discussion based on the Reproductive Life plan, including information about reproduction and a brochure with the same information.
  Arms: Intervention group

SUMMARY:
Many women and men are at risk for sexual transmitted infections and unwanted pregnancies and have unrealistic family planning intentions and insufficient knowledge of health promoting lifestyle prior to conception. Without sufficient support from the health care system this can lead to negative consequences. The aim of our study was to investigate if the usage of the Reproductive Life Plan in midwifery counselling increases women's knowledge of reproduction and particularly knowledge of folic acid intake prior to pregnancy. Secondary aims were to evaluate the influence on women's family planning and to further explore how women experienced the Reproductive Life Plan-based counselling.

ELIGIBILITY:
Inclusion Criteria:

* Visitor at the Student Health Clinic

Exclusion Criteria:

* Not speaking Swedish
* Male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Knowledge of reproduction | 2 months after the intervention
  Knowledge will be measured by knowledge of the following:
  * the fecundity of an ovum
  * how likely it is that a 25-year old women gets pregnant if she has unprotected intercourse at the time of ovulation
  * at what age there is a marked decline in women's ability to become pregnant
  * baby take home rate after IVF-treatment
  * factors that can impair female fertility
  * healthy lifestyle during pregnancy planning

SECONDARY OUTCOMES:
Family Planning Intentions | 2 months after the intervention
  Family planning intentions will be measured by the following questions:
  * Do you want (more) children in your life?
  * If yes, how many (more) children do you want?
  * If yes, at which age would you like to have your first/next child?
  * If yes, at which age you like to have your last child?

OTHER OUTCOMES:
Experience of the intervention | 2 months after the intervention
  Experience of the intervention is measure by
  * The overall experience of the intervention (very positive - very negative)
  * If the intervention made them think about reproduction in a different way
  * If the intervention made them search for more information about reproduction
  * The likelihood of approaching a midwife if they have more questions about reproduction
  * If they considered that midwifes or other health care professionals routinely should discuss the Reproductive Life Plan with their patients

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Stern, Principal Investigator — Uppsala University; Tanja Tydén, PhD, Study Director — Uppsala University; Margareta Larsson, PhD, Study Director — Uppsala University
Locations (1):
- The Student Health Centre, Uppsala, Sweden

REFERENCES:
- [Background] Moos MK. Unintended pregnancies: a call for nursing action. MCN Am J Matern Child Nurs. 2003 Jan-Feb;28(1):24-30; quiz 31. PMID 12514353
- [Background] Sanders LB. Reproductive life plans: initiating the dialogue with women. MCN Am J Matern Child Nurs. 2009 Nov-Dec;34(6):342-7; quiz 348-9. doi: 10.1097/01.NMC.0000363681.97443.c4. PMID 19901694
- [Background] Johnson K, Posner SF, Biermann J, Cordero JF, Atrash HK, Parker CS, Boulet S, Curtis MG; CDC/ATSDR Preconception Care Work Group; Select Panel on Preconception Care. Recommendations to improve preconception health and health care--United States. A report of the CDC/ATSDR Preconception Care Work Group and the Select Panel on Preconception Care. MMWR Recomm Rep. 2006 Apr 21;55(RR-6):1-23. PMID 16617292
- [Derived] Stern J, Larsson M, Kristiansson P, Tyden T. Introducing reproductive life plan-based information in contraceptive counselling: an RCT. Hum Reprod. 2013 Sep;28(9):2450-61. doi: 10.1093/humrep/det279. Epub 2013 Jul 10. PMID 23842564
- See also: Home page of Department of Public Health and Caring Sciences at Uppsala University — http://www.pubcare.uu.se/?languageId=1